CLINICAL TRIAL: NCT01581255
Title: The Effect of High Frequency Oscillation on Biological Markers of Lung Injury
Status: Terminated | Type: Observational
Why Stopped: Parent study (OSCILLATE) stopped by the Data Monitoring Committee
Sponsor: Canadian Critical Care Trials Group (Other)
Collaborators: Canadian Intensive Care Foundation (Other)
Responsible Party: Sponsor
Other Study IDs: OSCILLATE Biomarkers Study
Record Dates: First submitted 2012-04-17; First posted 2012-04-20 (Estimated); Last update posted 2012-09-12 (Estimated); Status verified 2012-09

CONDITIONS: Acute Respiratory Distress Syndrome
Keywords: acute respiratory distress syndrome; high frequency oscillation ventilation; ventilator-induced lung injury; biomarkers
MeSH Terms: conditions — Respiratory Distress Syndrome; Ventilator-Induced Lung Injury

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood samples will be drawn to measure the following biomarkers of ventilator-induced lung injury: IL-1β, IL-6, IL-8, IL-10, IFN-γ, TGF-β, TNF-α, VEGF, sICAM-1, surfactant protein D (SP-D), Krebs von den Lungen protein (KL-6), Clara cell 16 kD protein (CC16), Angiopoietin-1, Angiopoietin-2, and vWF.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Conventional lung protective ventilation: Critically-ill patients with the acute respiratory distress syndrome randomized to the conventional lung protective ventilation arm of the OSCILLATE trial.
- High frequency oscillation ventilation: Critically-ill patients with the acute respiratory distress syndrome randomized to the high frequency oscillation ventilation arm of the OSCILLATE trial.

SUMMARY:
Mechanical ventilation, although life-saving, damages the lungs through what is known as ventilator-induced lung injury. High frequency oscillation ventilation has been proposed as a ventilation method that may be less injurious to the lungs than conventional mechanical ventilation and may lead to better patient outcomes. To evaluate this hypothesis, the OSCILLATE trial is comparing outcomes in patients with the acute respiratory distress syndrome randomized to high frequency oscillation ventilation vs conventional lung protective ventilation. The present study is a substudy of the OSCILLATE trial looking at biomarkers of ventilator-induced lung injury in blood samples drawn from patients enrolled in OSCILLATE. The objective is to look for biochemical evidence of decreased ventilator-induced lung injury in patients treated with high frequency oscillation ventilation relative to conventional ventilation.

ELIGIBILITY:
Inclusion Criteria:

* enrollment in OSCILLATE (NCT01506401)

Exclusion Criteria:

* inability to provide blood samples

Ages: 16 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Critically-ill patients with the acute respiratory distress syndrome enrolled in the OSCILLATE trial (NCT01506401).
Sampling Method: Non-Probability Sample
Enrollment: 2 (Actual)
Dates: Start 2012-02; Primary Completion 2012-08 (Actual); Study Completion 2012-08 (Actual)

PRIMARY OUTCOMES:
Change from baseline in biomarkers of ventilator-induced lung injury | 24 hrs
  The following biomarkers will be measured in patients enrolled in both arms of the OSCILLATE trial (high frequency oscillation ventilation and conventional lung protective ventilation) at randomization and again at 24 hrs post randomization: IL-1β, IL-6, IL-8, IL-10, IFN-γ, TGF-β, TNF-α, VEGF, sICAM-1, surfactant protein D (SP-D), Krebs von den Lungen protein (KL-6), Clara cell 16 kD protein (CC16), Angiopoietin-1, Angiopoietin-2, and vWF.

CONTACTS AND LOCATIONS:
Overall Officials: Alexandra Binnie, MD, DPhil, Principal Investigator — University of Toronto; Claudia dos Santos, MD, PhD, Principal Investigator — University of Toronto; Niall Ferguson, MD, MSc, Principal Investigator — University of Toronto
Locations (2):
- Canada (2):
  - St Michael's Hospital, Toronto, Ontario
  - University Health Network, Toronto, Ontario

REFERENCES:
- See also: OSCILLATE trial — http://clinicaltrials.gov/ct2/show/NCT01506401